CLINICAL TRIAL: NCT00006375
Title: A Phase I Clinical and Pharmacokinetic Evaluation of LY293111 in Patients With Solid Tumors (Protocol H6H-MC-JEAI)
Brief Title: LY293111 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-076; CDR0000068249 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-H6H-MC-JEAI; NCI-G00-1862
Record Dates: First submitted 2000-10-04; First posted 2004-02-12 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — LY 293111

INTERVENTIONS:
Drug: LY293111

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of LY293111 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of LY293111 in patients with advanced solid tumors. II. Determine the safety profile and pharmacokinetics of this regimen in these patients. III. Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral LY293111 twice daily. Treatment continues for a maximum of 6 months in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of LY293111 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose limiting toxicity. Additional patients are treated at the MTD. Patients are followed at 30 days.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced and/or metastatic solid tumor for which no curative therapy exists No hematologic malignancies Measurable or evaluable disease No known CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) ALT and AST no greater than 2.0 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No concurrent systemic disorder that would preclude study No active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No concurrent immunotherapy Chemotherapy: No more than 3 prior chemotherapy regimens for metastatic disease At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered No other concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior anticancer hormonal therapy and recovered No concurrent anticancer hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: At least 4 weeks since prior investigational therapy No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York